CLINICAL TRIAL: NCT01905696
Title: The Role of S-nitrosohemoglobin in Regulating Systemic Blood Flow Under Hypoxic and Normoxic Conditions
Brief Title: The Role of S-nitrosohemoglobin in Regulating Systemic Blood Flow During Hypoxia and Normoxia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00041312
Record Dates: First submitted 2013-04-30; First posted 2013-07-23 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Focus is Determination of the Role of SNO-Hb in Forearm Blood Flow Regulation
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N-Acetylcysteine (NAC) (Experimental): After initial measurements of SNO-Hb level, forearm blood flow in response to exercise and hypoxia, subjects will take oral NAC 600 mg twice daily. Measurements will then be repeated.
  Interventions: Drug: Oral N-acetylcysteine

INTERVENTIONS:
Drug: Oral N-acetylcysteine

SUMMARY:
Nitric oxide is believed to contribute to regulation of blood flow by its selective binding to circulating hemoglobin (forming S-nitrosohemoglobin, SNO-Hb) and release in a PO2-dependent manner. This study is designed to test that hypothesis by measuring the effect of hypoxia and exercise on forearm blood flow before and after depletion of SNO-Hb using oral N-acetylcysteine.

DETAILED DESCRIPTION:
NO has been shown to associate with erythrocytes in the form of SNO-Hb and can deliver vasomotor changes as erythrocytes pass through a physiologic O2 gradient. The aim of this study is to transiently deplete circulating SNO-Hb levels to prove that these levels are directly linked with the normal physiological vasodilation that occurs in response to brief hypoxia that occurs in moderate exercise. This study will be performed on healthy volunteers especially with no predisposing cardiovascular or respiratory conditions that may change their vasomotor response to hypoxia. Systemic blood flow will be approximated using non-invasive forearm venous occlusion plethysmography which will be performed initial to gather baseline data. The participants will then undergo 4 days of 600 mg BID oral N-acetylcysteine (NAC) solution treatment which acts as a bait reactant for NO groups bound to hemoglobin (SNO-Hb) and will then undergo retesting with forearm plethysmography. At the time of both blood flow measurements, arterial blood samples will also be gathered via an arterial catheter inserted on each of two testing days to determine SNO-Hb levels. Statistical analysis will include measuring the blunting of the hypoxia response and SNO-Hb levels using baseline testing as a self-control for each participant. Large scale human placebo-controlled trials with high-dose oral NAC (up to 8000 mg/day) for periods up to 12 months have shown no clinically significant adverse reactions, much less than in the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Pregnancy
* smoking
* pulmonary disease
* cardiovascular disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States